CLINICAL TRIAL: NCT07266038
Title: Effectiveness of Cross K-wire Vs Lateral Entry K-wire Fixation in Maintaining Reduction of Gartland Type # Supracondylar Fractures of Children : A Comparative Study
Brief Title: Effectiveness of Cross K-wire Vs Lateral Entry K-wire Fixation in Maintaining Reduction of Gartland Type 3 Supracondylar Fractures of Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laiba Qamar (Other)
Collaborators: Bahawal Victoria Hospital Bahawalpur (Other)
Responsible Party: Sponsor-Investigator, Laiba Qamar, Principal Investigator, University of Health Sciences Lahore
Organization: University of Health Sciences Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #CVSLKWIRE3#
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Gartland Type 3 Supracondylar Fracture
Keywords: K-wire; supracondylar Frcature; Fixation; Loss of reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): The participants enrolled in this arm will be treated with cross K wire fixation
  Interventions: Procedure: Cross K Wire Fixation
- Group B (Experimental): The participants enrolled in this arm will be treated with lateral fixation of K wire after supracondylar fracture.
  Interventions: Procedure: Lateral K wire Fixation

INTERVENTIONS:
Procedure: Cross K Wire Fixation — In this intervention the K wire will be fixed in a Manner of Cross at the site of frature.
  Arms: Group A
Procedure: Lateral K wire Fixation — In this arm of intervention the K wire will be fixed laterally at the site of fracture.
  Arms: Group B

SUMMARY:
This study compares the efficacy of K wire when inserted in Cross V/s Lateral Direction in Supracondylar fractures of Gartland Type 3 in children. A comparative study.

DETAILED DESCRIPTION:
This is a randomized control trial being done to compare the efficacy of Cross V/S Laterally Placed K wire In Supracondylar fractures to calculate and copmpare the Post K wire iinsertion range of motion . It is also intended to calculate the frequency of loss of reduction after lateral K wire in terms of Skaggs Criteria . This study intends to find the better method of K wire fixatio to avoid the post fixation loss of reduction.

ELIGIBILITY:
Inclusion Criteria:

All male and female patients of age 02-13 years with Gartland type 3 Supracondylar Fracture of Humerus less than 7 days old

Exclusion Criteria:

patients with open fractures patients with neurovascular injuries patients with medial column communition Fractures more than 7 Days old Ipsilateral fractures of radius/ulna or shaft of humerus pathological fractures which are associated with bone density changes

Ages: 2 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
frequency of post K wire fixation loss of reduction | 2 months
  It is comonly noted that after lateral K wire fixation there is more frequent loss of reduction as compared to cross fixation method. The frequency of loss of reduction will be noted after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No